CLINICAL TRIAL: NCT04426019
Title: Using an Evidence-based Lay Health Worker Program to Increase Breast and Cervical Cancer Screening in Low-Income Hispanic Women in Houston
Brief Title: Using a Lay Health Worker Program to Increase Breast and Cervical Cancer Screening in Low-Income Hispanic Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas Health Science Center, Houston (Other)
Collaborators: Cancer Prevention Research Institute of Texas (Other)
Responsible Party: Principal Investigator, Lara Savas, Assistant Professor, The University of Texas Health Science Center, Houston
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: HSC-SPH-11-0179
Record Dates: First submitted 2020-05-27; First posted 2020-06-11 (Actual); Last update posted 2023-10-12 (Actual); Status verified 2023-10

CONDITIONS: Breast Cancer; Cervical Cancer
Keywords: Mammogram; Pap test
MeSH Terms: conditions — Breast Neoplasms; Uterine Cervical Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CLS intervention (Experimental): Community health workers (CHWs) assess women's breast and/or cervical cancer screening needs and deliver behavioral education designed to increase breast and/or cervical cancer screening. After completing the education, CHWs provide women with clinic referrals to local and affordable screening services. Participants also are offered telephone-delivered navigation support, which focuses on helping women overcome logistic and personal barriers to accessing screening services.
  Interventions: Behavioral: CLS Intervention
- No CLS intervention (Active Comparator): Community health workers (CHWs) assess women's breast and/or cervical cancer screening needs and deliver print materials to women describing cancer screening guidelines.
  Interventions: Behavioral: No CLS intervention

INTERVENTIONS:
Behavioral: CLS Intervention — Community health workers (or promotoras) will deliver the CLS program either in face-to-face and/or group sessions to all women within 2 months of the baseline interview. Each session will last approximately 1 to 2 hours, and will include CLS materials adapted for this study.At the conclusion of the CLS program, promotoras will provide information about local and affordable providers delivering low-cost or free breast and cervical cancer screening services. Should a woman require follow-up for abnormal results, referrals will be given to programs,which provides assistance accessing cancer diagnostic and treatment services. Two weeks after delivering the education component of the CLS program, promotoras will call women to provide any further assistance needed. During these follow-up calls promotoras will provide on-going navigation support to women in need of mammography and Pap test screening
  Other Names: CHW-delivered education
  Arms: CLS intervention
Behavioral: No CLS intervention — This control arm will receive only usual practice care (print education) and will not receive the CLS intervention. They may receive the intervention after the study has been completed
  Other Names: Usual Care
  Arms: No CLS intervention

SUMMARY:
The primary purpose of this study is adapt the Cultivando la Salud (CLS) intervention for a new community and priority population and to train community health workers (promotoras) from the Prosalud promotora program to implement the adapted CLS breast and cervical cancer screening program. The adaptation and delivery of the CLS intervention program focuses on meeting the needs and supporting of CHWs and Hispanic/Latina women in the Greater Houston Area. Finally, this study aims to evaluate the process and effect of the adapted CLS program (renamed Salud en Mis Manos (SEMM) on increasing mammography and cervical cancer screening.

DETAILED DESCRIPTION:
CHWs identify women in the community in need of breast and/or cervical cancer screening. Based on their screening needs, they invite women to participate in the CLS behavioral intervention. Women are randomized to intervention and usual care comparison (delayed intervention) groups. After women are consented to participate in the study, the study team administers the baseline survey. After the baseline survey is administered, the CLS-adapted intervention (renamed Salud en Mis Manos), is delivered to participants randomized to the intervention group. After the follow-up survey is administered to the participants, women in the comparison group are offered the CLS (SEMM) intervention.

ELIGIBILITY:
Inclusion Criteria:

* women who identify as Hispanic/Latina ancestry or descent and live in the Greater Houston Area in Texas
* no previous diagnosis of breast or cervical cancer

Exclusion Criteria:

* Pregnant women, and women who are adherent to screening guidelines
* prior or current cancer diagnosis

Min Age: 21 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1025 (Actual)
Dates: Start 2012-01-12 (Actual); Primary Completion 2014-05-16 (Actual); Study Completion 2014-05-16 (Actual)

PRIMARY OUTCOMES:
The primary outcome for breast cancer screening outcome based on mammography screening behavior measured among participants using self-report. | end of evaluation period (6 month follow-up survey, through completion of hard to follow-up period on average 10 months).
  Outcomes based on self-report on follow-up survey
The primary outcome for cervical cancer screening outcome based on Pap screening behavior measured among participants using self-report. | end of evaluation period (6 month follow-up survey, through completion of hard to follow-up period on average 10 months).
  Outcomes based on self-report on follow-up survey

CONTACTS AND LOCATIONS:
Overall Officials: Lara Savas, Principal Investigator — The University of Texas Health Science Center, Houston
Locations (1):
- The University of Texas Health Science Center at Houston, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No